CLINICAL TRIAL: NCT02217033
Title: A Pilot Study Evaluating the Effect of 'R' (Electro-Kinetically Altered Beverage) on Insomnia, Fatigue and Depression in Breast Cancer Patients Receiving Adjuvant Chemotherapy
Brief Title: Effects of 'R' (Electro-kinetic Beverage) on Insomnia, Fatigue, and Depression in Breast Cancer Patients Having Adjuvant Chemo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After an interim analysis the Company providing the product decided not to continue with the study
Sponsor: South Sound Care Foundation (Other)
Responsible Party: Principal Investigator, Francis (Frank) Senecal, MD, Site Principal Investigator, South Sound Care Foundation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: R822662
Record Dates: First submitted 2014-08-08; First posted 2014-08-15 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Stage I breast cancer; Stage II breast cancer; Water study; 'R'; Electro-kinetically altered beverage; altered beverage; Insomnia; Fatigue; Depression; Adjuvant chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders; Fatigue; Depression | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purified Water (Placebo Comparator): In this arm, eligible subjects will begin to consume purified water (placebo) just prior to the 1st cycle of chemotherapy. Subjects will continue to consume the placebo through their chemotherapy and then for an additional 12 weeks after completing chemotherapy.
  Subjects will consume a specific volume based on the following weight categories: <150 lb = 2 bottles/day; ≥150 lb and <225 lb = 3 bottles/day; ≥225 lb = 4 bottles/day. Subjects will consume placebo for a minimum of 168 days.
  Interventions: Other: Placebo (water)
- 'R' (Electro-kinetically altered beverage) (Experimental): Patients randomized to this arm will begin to consume "R" (Electro-kinetically altered beverage) just prior to the 1st cycle of chemotherapy and continue it through their chemotherapy cycles and then for an additional 12 weeks after completing chemotherapy.
  Subjects will consume a specific volume based on the following weight categories: <150 lb = 2 bottles/day; ≥150 lb and <225 lb = 3 bottles/day; ≥225 lb = 4 bottles/day. Subjects will consume R for a minimum of 168 days.
  Interventions: Other: 'R' (Electro-kinetically altered beverage)

INTERVENTIONS:
Other: 'R' (Electro-kinetically altered beverage)
  Arms: 'R' (Electro-kinetically altered beverage)
Other: Placebo (water)
  Arms: Purified Water

SUMMARY:
The purpose of this study is to evaluate the effects of consuming "R" on quality of life in the areas of insomnia, fatigue, and depression in female breast cancer patients receiving multi-cycle adjuvant chemotherapy.

DETAILED DESCRIPTION:
Female breast cancer patients eligible for adjuvant therapy with four cycles of Taxotere and Cytoxan chemotherapy after surgery will be enrolled for the study.

Eligible subjects will begin to consume either "R" or purified water (placebo) just prior to the 1st cycle of chemotherapy. Subjects will continue to consume either "R" or placebo through Cycle 1, Cycle 2, Cycle 3, Cycle 4, and for an additional 12 weeks after completing chemotherapy.

Study procedures will include clinical lab assessments, analysis of inflammatory markers, RNA biomarkers, adverse events, subject diary, and quality of life measurements for insomnia, fatigue and depression.

ELIGIBILITY:
Inclusion Criteria:

* Female, non-smokers ≥ 18 years of age
* Histologically or cytologically confirmed diagnosis of Stage I or II adenocarcinoma of the breast and a candidate for adjuvant chemotherapy
* Scheduled to receive 4 cycles of adjuvant Taxotere and Cytoxan chemotherapy (TC): docetaxel 75 mg/m2 and cyclophosphamide 600 mg/m2 administered intravenously on Day 1 of each 21-day cycle
* Eastern Cooperative Oncology Group Status (ECOG) performance status of ≤ 1
* No prior treatment for breast cancer other than surgery
* Adequate baseline organ function as evidenced by:

  * Hemoglobin ≥ 9 g/dL
  * Absolute neutrophil count ≥ 1.5 x 109 cells/mm3
  * Platelet count ≥ 100,000 cells/mm3
  * Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
  * Alkaline phosphatase ≤ 1.5 x ULN
* No history of other malignancies within the last 5 years, except for carcinoma in situ of the cervix, or basal cell carcinoma or squamous cell carcinoma of the skin that have been previously treated with curative intent
* Women of childbearing potential who commit to using two forms of highly effective non-hormonal contraception either by the subject and/or partner during the study
* Negative urine pregnancy test at screening
* Negative urine drug screen (UDS) for drugs of abuse including cotinine (nicotine) at screening
* Subjects must be capable of understanding the purpose and risks of the study and provide written, voluntary informed consent

Exclusion Criteria:

* Preexisting diagnosed psychiatric disorder as defined by The Diagnostic and Statistical Manual (DSM) of Mental Disorders (published by the American Psychiatric Association). Subjects with a diagnosis of depression will be allowed to enter into study as long as they have been treated with medication for ≥ 6 months and/or depression is considered to be well controlled
* Pregnant or lactating
* Diabetes
* Concomitant use of any sleeping agents during the course of the study (Anti- anxiety medications will be allowed)
* Steroid therapy other than the standard prescribed therapy of either of the following during the course of the study:

  * Dexamethasone 4-12 mg IV on Day 1 of any cycle
  * Dexamethasone 4-12 mg PO on Day 2 and Day 3 of any cycle
* Anti-estrogen therapy other than the standard prescribed therapy of one of the following:

  * Tamoxifen/Nolvadex 20 mg PO daily
  * Anastrazole/Arimidex 1 mg PO daily
  * Letrozole/Femara 2.5 mg PO daily
  * Exemestane/Aromasin 25 mg PO daily
* Use of any other antiemetic regimen other than the following (with the exception of PO antiemetics):

  * Emend /Aprepitant150 mg IV on Day 1 of any cycle
  * Aloxi/Palonosetron 0.25 mg IV on Day 1 of any cycle
  * Dexamethasone 8 mg IV on Day 1 of any cycle
  * Dexamethasone 8 mg PO on Day 2 and Day 3 of any cycle
  * Zofran/Ondansetron 12 mg IV on Day 1 of any cycle
  * Kytrile/Granisetron 1-2 mg IV on Day 1 of any cycle
* Therapy with any immunomodulatory or immunosuppressive drugs within 6 months prior to enrollment
* Known history of positive viral serology test for Human Immunodeficiency Virus (HIV-1), HBsAG and Hepatitis C antibody
* Any change in the initially prescribed chemotherapy
* Use of herbal remedies, dietary supplements or mega-vitamins, with the exception of a multi-vitamin
* Investigator deems the subject to be unable or unwilling to comply with the requirements of the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The effects of consuming "R" on quality of life in the areas of insomnia in breast cancer patients receiving multi-cycle adjuvant chemotherapy | Patients will be followed for up to 25 weeks
  SleepMed Insomnia Questionnaire: This is a test to assess, in general, how a subject is feeling about their sleep using a "0-4" point scale - with the "0" representing no problem with sleep and "4" representing a big problem with how a subject feels about the quality of their sleep.
The effects of consuming "R" on quality of life in the areas of fatigue in breast cancer patients receiving multi-cycle adjuvant chemotherapy | Patients will be followed for up to 25 weeks
  FACIT Fatigue Scale: A list of questions that asks a patient how fatigued they have felt in the last 7 days.

SECONDARY OUTCOMES:
The effects of consuming "R" on quality of life in the areas of depression in breast cancer patients receiving multi-cycle adjuvant chemotherapy | Patients will be followed for up to 25 weeks
  Beck Depression Inventory-II: A list of statements that ask a subject about the way they have been feeling for the last two weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Francis (Frank) Senecal, MD, Principal Investigator — Northwest Medical Specialties
Locations (6):
- United States (6):
  - NWMS Bonney Lake - Medical Oncology, Bonney Lake, Washington
  - NWMS Federal Way - Medical Oncology, Federal Way, Washington
  - NWMS Gig Harbor - Medical Oncology, Gig Harbor, Washington
  - NWMS Lakewood - Medical Oncology, Lakewood, Washington
  - Rainier Hematology-Oncology, WA, Puyallup, Washington
  - NWMS Tacoma - Medical Oncology & Infectious Diseases, Tacoma, Washington